CLINICAL TRIAL: NCT02518737
Title: Examination of the Postprandial Bone Remodeling in Persons With Reduced Activity of the Receptor for the Enteric Hormone Glucose-dependent Insulinotropic Polypeptide
Brief Title: Examination of the Postprandial Bone Remodeling in Persons With Reduced GIP-Receptor Activity
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Bolette Hartmann, PhD, Associate Professor, University of Copenhagen
Other Study IDs: GRD
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Bone Remodeling
Keywords: Glucose-dependent Insulinotropic Polypeptide; Receptor Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GIP-receptor deficient: Persons with a mutation (Glu354Gln) causing their GIP-receptor to loose function.
  Interventions: Other: Meal Test
- Controls: Matched controls, with a normal functioning GIP-receptor.
  Interventions: Other: Meal Test

INTERVENTIONS:
Other: Meal Test

SUMMARY:
The bone tissue of the human adult body is in a constant process of break-down (resorption) and rebuilding (formation), a process called bone remodeling. The extent to which bone remodeling happens varies during the day, especially a decrease in the bone resorption is observed after eating.

The overall purpose of this study is to examine the possible role of the hormone Glucose-dependent Insulinotropic Polypeptide (GIP) in Bone Remodeling. GIP is released from cells in the gut after eating, and previous studies have shown an effect of GIP on bone tissue. In addition, it has been observed that the risk of bone fracture is 60% higher in women with a mutation in the GIP receptor, when compared to women with a normal functioning GIP receptor.

In the present study humans with a mutation in their GIP receptor is compared to humans with a normal functioning GIP receptor. The study population will be examined during a meal stimulation test, where blood will be sampled regularly. The blood samples will be examined for markers of bone resorption among other markers of bone remodeling, GIP and other gut hormones.

The hypothesis for the present study is that GIP secreted after meal ingestion inhibits bone resorption. Thus it is expected that the decrease in resorption is less pronounced in the humans carrying the GIP-receptor mutation, compared to humans with a normal functioning GIP receptor.

ELIGIBILITY:
Inclusion Criteria:

* Verified mutation (Glu354Gln) of the GIP-receptor

Exclusion Criteria:

* Type 2 diabetes
* Pregnancy
* Previous long-lasting treatment with steroids
* On-going steroid treatment (with the exception of inhalation-steroids)
* Osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups will be recruited from the Helbred2006 cohort, Glostrup Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
CTx | 7, 15, 30, 45, 60, 90, 120, 150, 180, 240 minutes after intake of the meal test.
  CTx is a biomarker of bone resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Bolette Hartmann, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Biomedical Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Qvist P, Christgau S, Pedersen BJ, Schlemmer A, Christiansen C. Circadian variation in the serum concentration of C-terminal telopeptide of type I collagen (serum CTx): effects of gender, age, menopausal status, posture, daylight, serum cortisol, and fasting. Bone. 2002 Jul;31(1):57-61. doi: 10.1016/s8756-3282(02)00791-3. PMID 12110413
- [Background] Nielsen HK, Brixen K, Kassem M, Christensen SE, Mosekilde L. Diurnal rhythm in serum osteocalcin: relation with sleep, growth hormone, and PTH(1-84). Calcif Tissue Int. 1991 Dec;49(6):373-7. doi: 10.1007/BF02555845. PMID 1818760
- [Background] Nissen A, Christensen M, Knop FK, Vilsboll T, Holst JJ, Hartmann B. Glucose-dependent insulinotropic polypeptide inhibits bone resorption in humans. J Clin Endocrinol Metab. 2014 Nov;99(11):E2325-9. doi: 10.1210/jc.2014-2547. Epub 2014 Aug 21. PMID 25144635
- [Background] Torekov SS, Harslof T, Rejnmark L, Eiken P, Jensen JB, Herman AP, Hansen T, Pedersen O, Holst JJ, Langdahl BL. A functional amino acid substitution in the glucose-dependent insulinotropic polypeptide receptor (GIPR) gene is associated with lower bone mineral density and increased fracture risk. J Clin Endocrinol Metab. 2014 Apr;99(4):E729-33. doi: 10.1210/jc.2013-3766. Epub 2014 Jan 21. PMID 24446656